CLINICAL TRIAL: NCT07384507
Title: Evaluation of Perioperative Recovery With a Spontaneous Breathing-Preserving Strategy in Older Lung Transplant Recipients: A Prospective Multicenter Single-Arm Cohort Study
Brief Title: Perioperative Recovery Outcomes With a Spontaneous Breathing Strategy in Older Lung Transplant Recipients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Chief Physician and Professor of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BREATH-Elderly
Record Dates: First submitted 2026-01-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: End-stage Lung Disease
Keywords: Lung transplantation; Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tubeless LTx Group (Experimental): All participants receive lung transplantation under a standardized spontaneous-breathing-preserving ("tubeless") pathway. After anesthesia induction, a supraglottic airway (laryngeal mask airway) is used when feasible with regional nerve blocks and multimodal sedation/analgesia to control pain and cough while maintaining spontaneous breathing. Muscle relaxants are minimized; ventilatory assistance is provided only as needed with low airway pressures. Postoperatively, patients are managed in the intensive care unit with spontaneous breathing and protocol-guided noninvasive respiratory support. Conversion to endotracheal intubation, invasive mechanical ventilation, and/or extracorporeal membrane oxygenation is allowed if predefined safety criteria are met.
  Interventions: Procedure: Lung transplantation that preserves spontaneous breathing function

INTERVENTIONS:
Procedure: Lung transplantation that preserves spontaneous breathing function — This intervention uses a spontaneous-breathing-preserving anesthesia strategy during lung transplantation, which differs from conventional management based on endotracheal intubation and invasive mechanical ventilation. A supraglottic airway (laryngeal mask airway) is used when feasible instead of endotracheal intubation to maintain spontaneous breathing throughout the procedure. Neuromuscular blocking agents are minimized, and regional nerve blocks (such as intercostal nerve blocks or paravertebral blocks) are used to control pain and suppress cough while preserving the patient's ability to breathe independently. After surgery, patients receive protocol-guided noninvasive respiratory support (for example, high-flow nasal oxygen or noninvasive ventilation), with the goal of avoiding routine invasive mechanical ventilation.

SUMMARY:
The goal of this prospective, multicenter, single-arm cohort study is to learn whether a lung transplantation approach that preserves patients' spontaneous breathing during surgery can improve early recovery in adults aged 70 years and older undergoing allogeneic lung transplantation.

The main questions it aims to answer are whether, in adult lung transplant recipients aged 70 years and older, an anesthesia-surgical strategy designed to preserve spontaneous breathing is associated with better early postoperative recovery, specifically in terms of the need for postoperative invasive mechanical ventilation, postoperative length of hospital stay, and perioperative survival.

Participants will undergo lung transplantation using a standardized anesthesia-surgical strategy intended to preserve spontaneous breathing, with predefined criteria for conversion to tracheal intubation and/or ECMO if clinically needed. They will receive standardized perioperative management and routine postoperative care (including ICU monitoring, rehabilitation, and recovery support) as determined by the transplant team. Participants will be assessed throughout hospitalization and followed for postoperative complications and outcomes through discharge and up to 30 days after surgery.

DETAILED DESCRIPTION:
This prospective, multicenter, single-arm cohort study (BREATH-Elderly) is designed to evaluate the clinical effectiveness and safety of an anesthesia-surgical strategy intended to preserve spontaneous breathing in adult lung transplant recipients aged 70 years and older. The primary objective is to characterize early postoperative recovery under this standardized pathway, with a focus on (1) postoperative invasive mechanical ventilation (IMV) requirement, (2) postoperative length of hospital stay (LOS), and (3) perioperative survival (from the start of transplantation to hospital discharge or postoperative day 30, whichever occurs first).

Eligible participants are adults aged ≥70 years who are listed for allogeneic lung transplantation and meet prespecified perioperative safety thresholds (e.g., not receiving ongoing invasive mechanical ventilation or ECMO preoperatively; acceptable baseline cardiac and renal function; no evidence of active infection; and adequate rehabilitation potential and caregiver support). Key exclusions include retransplantation or multi-organ transplantation, recent major cardiovascular/cerebrovascular events, severe end-organ failure, active malignancy, extreme body habitus (e.g., BMI <16 or ≥35 kg/m²), ongoing substance use, and scenarios judged by the anesthesia team to make a preserved spontaneous-breathing pathway unsafe (e.g., predicted difficult airway or inability to safely manage the airway with a laryngeal mask-based approach).

All enrolled participants will undergo lung transplantation using a standardized preserved spontaneous-breathing anesthesia-surgical pathway, typically based on total intravenous anesthesia with airway management using a laryngeal mask airway and continuous monitoring of oxygenation and ventilation. The protocol includes predefined rescue escalation criteria and standardized procedures for conversion when clinically indicated. Triggers for conversion may include, but are not limited to: persistent hypoxemia (e.g., SpO₂ <85% despite assisted ventilation), severe hypercapnia with acidosis and accompanying hemodynamic/arrhythmic instability (e.g., PaCO₂ ≥80 mmHg with repeated pH <7.25 and circulatory/arrhythmic changes), unstable surgical field due to marked mediastinal movement refractory to adjustment, major intraoperative bleeding impairing operative safety, and abnormal airway secretions (e.g., increased or bloody sputum with a >30% reduction in tidal volume or elevated airway pressure when assisted ventilation is required). If conversion is required, the protocol specifies intubation approach options (e.g., single-lumen tube plus bronchial blocker or double-lumen tube when lung isolation is necessary) and immediate initiation of lung-protective ventilation. Postoperative care, including immunosuppression and infection prevention, follows routine standards at each participating transplant center and is recorded in the case report form. Participants are assessed throughout the index hospitalization, with key postoperative complications captured through discharge and up to 30 days after surgery, and additional follow-up items (e.g., 90-day survival/readmission/interventions) recorded where applicable.

The primary endpoint is a composite of three early recovery indicators (reported both as a composite and as individual components): (1) postoperative IMV requirement in the early postoperative period (including events such as re-intubation/tracheostomy and/or new or escalated extracorporeal respiratory support as defined in the protocol), (2) postoperative LOS, and (3) perioperative survival to discharge or postoperative day 30. Secondary endpoints include intraoperative and anesthesia-related measures (e.g., operative/anesthesia time, blood loss, perioperative medication exposure, success rate of removing the airway device in the operating room, time to first effective communication), ICU length of stay, in-hospital resource utilization/cost categories, and a prespecified list of postoperative complications (e.g., primary graft dysfunction graded at standard time points, respiratory support escalation events, infections, bleeding requiring re-intervention, AKI and renal replacement therapy, major cardiovascular/cerebrovascular events, rejection episodes, and thrombotic events). Outcomes will be summarized descriptively and compared against each center's historical outcomes under conventional intubated strategies using appropriate one-sample methods; multivariable models may be used to adjust for important clinical factors (e.g., diagnosis, intraoperative ECMO use, and procedural complexity) when warranted.

The study is expected to demonstrate that, in carefully selected recipients aged ≥70 years, a standardized preserved spontaneous-breathing strategy is feasible and can be implemented with structured rescue pathways, and may be associated with a higher proportion of patients avoiding postoperative IMV, a shorter postoperative hospital stay, and maintained perioperative survival within an acceptable safety profile. These findings are intended to support broader implementation guidance and inform the design of subsequent comparative studies in elderly lung transplant populations.

ELIGIBILITY:
[1] Inclusion Criteria

1. Age and informed consent: Age ≥70 years; able to understand the study and provide written informed consent, or, where permitted by ethics and applicable regulations, consent may be provided by a legally authorized representative (LAR)/authorized surrogate; willing and able to complete follow-up.
2. Transplant candidacy: Listed in CLuTR or the lung transplant waiting list of the participating center, with a plan to undergo allogeneic lung transplantation.
3. Preoperative support status: Not receiving ongoing invasive mechanical ventilation (endotracheal intubation or tracheostomy) preoperatively, and not receiving ECMO or other extracorporeal life support.
4. Minimum key organ function: LVEF ≥40%; eGFR ≥40 mL/min/1.73 m²; no evidence of acute liver failure or decompensated cirrhosis/portal hypertension; ASA physical status ≤ IV (American Society of Anesthesiologists classification).
5. Infection and communicable diseases: No evidence of active infection; no active tuberculosis; HIV/HBV/HCV status meets the center's transplant requirements (e.g., undetectable viral load, as applicable).
6. Rehabilitation and support: Demonstrated potential for postoperative rehabilitation (able to participate in training) and reliable caregiving support (at least one primary caregiver).

[2] Exclusion Criteria

1. Informed consent/adherence: Refusal or withdrawal of informed consent; investigator judgment that follow-up cannot be completed or there is recurrent severe non-adherence.
2. Transplant type: Re-transplantation, multi-organ transplantation, or planned lobar lung transplantation.
3. Recent major cardio-cerebrovascular events: Acute coronary syndrome/myocardial infarction or stroke within the past 30 days.
4. Severe organ dysfunction/acute failure: LVEF <40%; eGFR <40 mL/min/1.73 m²; acute liver failure or decompensated cirrhosis/portal hypertension; acute renal failure requiring dialysis with low likelihood of recovery; significant preoperative neuropsychiatric disorders or altered consciousness.
5. High risk of severe infection: Septic shock; active extrapulmonary/disseminated infection; active tuberculosis; detectable HIV viral load (or otherwise not meeting the center's transplant criteria).
6. High bleeding risk: Severe bronchiectasis without preoperative vascular intervention or not correctable/mitigable.
7. Malignancy: Active malignancy or tumors with high risk of recurrence or high cancer-related mortality risk.
8. Extreme body habitus/major deformity: BMI ≥35 kg/m² or BMI <16 kg/m²; clearly diagnosed severe chest wall deformity or spinal deformity.
9. Substance use/dependence: Current use of cigarettes, e-cigarettes, smoked/vaped cannabis, or intravenous drug use.
10. Tubeless/spontaneous-breathing strategy not safely feasible: Deemed by the anesthesia team to have a difficult airway or unsafe supraglottic/non-intubated airway management (e.g., anticipated intraoperative airway difficulty, pharyngeal/laryngeal stenosis not suitable for a laryngeal mask), including but not limited to: Mallampati class >III, mouth opening <3 cm, thyromental distance <5 cm, or significant airway anatomical variations (e.g., aberrant right upper lobe bronchial takeoff with planned right lung transplantation) where safe management with LMA/single-lumen approaches is judged unlikely.
11. Donor/donor lung limitations: Donor age >60 years; donor mechanical ventilation >14 days; positive donor airway microbiology considered unacceptable by the transplant team.
12. Protected populations: Pregnant or breastfeeding women.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Requiring Postoperative Invasive Mechanical Ventilation (IMV) During Index Hospitalization | From ICU admission immediately after leaving the operating room until hospital discharge or in-hospital death, assessed up to 90 days postoperatively (if hospitalization extends beyond 90 days, events after day 90 will not be counted for this outcome).
  Number of participants who require postoperative invasive mechanical ventilation (IMV) delivered via an endotracheal tube or tracheostomy tube at any time after leaving the operating room and before hospital discharge (including in-hospital death).
Postoperative Hospital Length of Stay (Days) During Index Hospitalization | From end of surgery (postoperative Day 0) until hospital discharge or in-hospital death (index hospitalization), assessed up to 90 days.
  The number of days from the end of surgery (postoperative Day 0) to the date the participant is discharged from the index hospitalization, according to institutional discharge criteria. Participants who die in hospital will be assigned length of stay through the date of in-hospital death.
Rate of Perioperative Survival | From start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first.
  Perioperative survival is defined as the proportion of participants who remain alive from the start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first. Participants who die before discharge or before postoperative Day 30 will be counted as non-survivors for this outcome.

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data (IPD) underlying the analyses of this clinical study, limited to baseline and perioperative variables. Baseline IPD will include demographics (e.g., age, sex), primary diagnosis, key comorbidities, and transplant-relevant preoperative measures and donor/recipient characteristics recorded in structured fields. Perioperative IPD will include operative and anesthesia strategy, airway management, intraoperative/early postoperative respiratory and hemodynamic parameters, major perioperative interventions (e.g., ECMO use), and key in-hospital outcomes during the index hospitalization (e.g., need for postoperative IMV, complications, ICU/hospital length of stay, and in-hospital mortality). The study protocol and statistical analysis plan will also be shared. All direct identifiers will be removed and dates will be shifted/aggregated as needed to protect privacy.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning at study completion and ending 2 years after study completion.
Access Criteria: De-identified IPD and supporting documents (study protocol, statistical analysis plan, and data dictionary) will be available to qualified researchers outside the primary study group for scientifically sound research purposes. Access will be granted upon submission of a written request that includes a brief research proposal, analysis plan, and proof of relevant ethics/IRB review if applicable. Requests will be reviewed by the study steering committee/data access committee. Approved requestors must sign a data use agreement prohibiting re-identification attempts and onward sharing, and requiring appropriate data security measures and acknowledgement of the original study. Data will be provided through a secure electronic transfer or a controlled-access online repository; access instructions will be provided after approval.
URL: https://www.gyfyyy.cn/